CLINICAL TRIAL: NCT05785416
Title: Effects of Proprioceptive Neuromuscular Facilitation on Joint Range of Motion, Flexibility and Electromyographic Activity of Knee Muscles in Older Adults
Brief Title: Stretching Techniques of Knee Muscles and Their Effect on Joint Range, Suppleness and Muscle Activity in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deepak Malhotra (Other)
Collaborators: Jamia Millia Islamia (Other)
Responsible Party: Sponsor-Investigator, Deepak Malhotra, Assistant Professor, Jamia Hamdard University
Organization: Jamia Hamdard University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16/9/121/JMI/IEC/2017
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Muscle Tightness; Muscle Weakness
Keywords: Contract Relax; Proprioceptive Neuromuscular Facilitation; Electromyography; Elderly; Flexibility; Range of Motion
MeSH Terms: conditions — Muscle Weakness | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: 30 males aged 55-75 years were randomly assigned into 3 arms - PNF group (n=10), Static Stretch group (n=10) and Control group (n=10)
Who Masked: Outcomes Assessor
Masking Description: outcome assessor-blinded pre-test post-test randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNF- CR Group (Experimental): The participants in the group were given PNF contract- relax stretching using the standard protocol. One trial had two isometric contractions each followed by five seconds muscle stretch and there was a total of four trials. Total of 12 sessions in 4 weeks (3sessions/week).
  Interventions: Other: Proprioceptive Neuromuscular Stretching - Contract Relax stretching (PNF-CR)
- Static Stretching Group (Experimental): The participants in the group were given sustained stretching for a period of 80s at a stretch.
  Total of 12 sessions in 4 weeks (3sessions/week).
  Interventions: Other: Static Stretching (SS)
- Control Group (No Intervention): No intervention was given in this group

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Stretching - Contract Relax stretching (PNF-CR) — PNF-CR utilized the concept of autogenic inhibition of the muscle for improving the flexibility of the muscle. It includes stretching a muscle after a brief period of activation.
  Arms: PNF- CR Group
Other: Static Stretching (SS) — The SS technique utilized the concept of creep for improving the hamstring flexibility. The stretch was maintained for a prolonged period passively by the therapist.
  Arms: Static Stretching Group

SUMMARY:
The goal of this clinical trial was to compare the effect of two different types of stretching techniques in elderly population. The main questions it aims to answer are:

1. What is the immediate effect (after a single intervention) of these stretching techniques on muscle flexibility, amount of knee joint motion and muscle activity?
2. What is the effect of a four week intervention program of these stretching techniques on muscle flexibility, amount of knee joint motion and muscle activity? There were three groups with ten randomly allocated participants in each group. Intervention group I was given a stretching technique called contract-relax technique and the Intervention group II was given static stretching. The third group was not given any treatment and was taken as a control. The main aim was to find out that whether the two techniques are effective or not and which one of the two is better than the other in terms of improvement in the above mentioned parameters.

DETAILED DESCRIPTION:
The objective of the study was to compare the effects of Proprioceptive Neuromuscular Facilitation - Contract Relax (PNF- CR) and static stretch techniques immediately and post four weeks of intervention on knee range of motion, flexibility and electromyographic activity of knee muscles among older adults. This is an outcome assessor-blinded pre-test post-test randomized controlled trial with two experimental groups (PNF-CR and Static Stretching) and a control group. 30 males aged 55-75 years were randomly assigned into PNF group (n=10), Static Stretch group (n=10) and Control group (n=10). Knee range of motion, electromyographic activity of hamstrings and sit and reach test, were taken for the dominant side thrice: pre-intervention, immediately after stretching and after the training period. Active knee range of motion (ROM) was assessed using a universal goniometer. Surface Electromyography (EMG) was used to record Maximal voluntary isometric contraction (MVIC) of biceps femoris and the Chair Sit-and-Reach Test (CART) was used to assess the hamstring muscle's length flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged between 55 and 75 years
* Able to do activities of daily living (ADL) without assistance
* Able to comprehend and follow instructions

Exclusion Criteria:

* Grade III or IV osteoarthritis or any other musculoskeletal condition affecting the muscle length.
* History of any surgery to hip, knee, low back or ankle
* History of any medication (anti-inflammatory, for pain relief, or anti-arthritic) in previous six months
* History of life-threatening disease (neurological disease, cardiovascular disease, severe hypertension)
* Passive full knee extension (popliteal angle 180 degrees)

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male participants were included in the study.
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Active Knee Range of Motion | Baseline, After 1st intervention (immediate), 4 weeks after intervention
  The active extension knee range of motion was measured using a universal goniometer.
Change in Maximum Voluntary Isometric Contraction (MVIC) | Baseline, After 1st intervention (immediate), 4 weeks after intervention
  The Electromyographic activity of the biceps femoris muscle was evaluated using the surface electrodes during the maximal isometric contraction.

SECONDARY OUTCOMES:
Change in Hamstring flexibility | Baseline, After 1st intervention (immediate), 4 weeks after intervention
  The hamstring flexibility was measured using the Chair Sit and Reach Test (CART)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Zaidi, MPT, Principal Investigator — Jamia Millia Islamia
Locations (1):
- Out Patient Department, Centre for Physiotherapy & Rehabilitation Sciences, Jamia Millia Islamia, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No